CLINICAL TRIAL: NCT06301347
Title: Integrated Parenting Intervention for Parents With Schizophrenia: A Feasibility Randomized Controlled Trial in Pakistan
Brief Title: Learning Through Play Plus for Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LTP+P
Record Dates: First submitted 2024-03-02; First posted 2024-03-08 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of the two treatment conditions (LTP Plus or TAU) through computer generated algorithm.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Learning through Play Plus (Experimental): The proposed intervention is a combination of two interventions:
  Learning through Play The 'Learning through Play' programme is intended to stimulate early child development. The central feature of the program is a pictorial calendar devised for parents, depicting eight successive stages of child development from birth to 3 years, with illustrations of parent-child play and other activities that promote parental involvement, learning, and attachment.
  Culturally Adapted Cognitive Behavioral Therapy for Psychosis (CaCBTp) The CaCBTp interventions will follow the treatment manual developed by David Kingdom and David Tarkington and culturally adapted by Farooq Naeem. In CBT the general approach will be a collaborative understanding of the development of symptoms and further work toward reducing distress and disability in participants.
  Interventions: Behavioral: Learning through Play Plus
- Treatment-as-Usual (No Intervention): This group of patients will not be provided any intervention. They will be taking only treament as usual (which in Pakistan means attending the outpatient clinic at regular intervals and taking prescribed medication) and we will compare this group with LTP Plus group after three months.

INTERVENTIONS:
Behavioral: Learning through Play Plus — Combination of two interventions: Learning through Play and Cognitive Behaviour Therapy
  Arms: Learning through Play Plus

SUMMARY:
Evidence reports that parents with schizophrenia are particularly vulnerable to parenting difficulties and also experience problems in sensitively interacting with their children. This may cause insecure attachment in infants of mothers with psychosis. Children of parents with schizophrenia have poor developmental and clinical outcomes. However, there is no published trial, to the best of our knowledge, for children of parents with schizophrenia. Learning through Play (LTP) is a potentially low cost intervention to improve maternal mental health and child outcomes by promoting health child development. The proposed study will integrate LTP with existing culturally appropriate Cognitive Behaviour Theray (CBT) for psychosis (CaCBT-p) and test its feasibility and acceptability for parents with schizophrenia.

DETAILED DESCRIPTION:
Objectives

* To determine whether the proposed intervention is acceptable to the parents with schizophrenia.
* To assess the feasibility of proposed intervention for target population (no of sessions attended, content, duration and location, uptake and retention).
* To determine most suitable outcome measures for future randomized controlled trial.
* To identify any barriers in recruitment of participants. Recruiting up to 75% of total sample will be a success criteria.

Methods Design: Mixed method feasibility Randomised Controlled Trial Study Sites The participants will be recruited from outpatient departments of psychiatry and community settings in 7 cities of Pakistan i.e. Karachi, Hyderabad, Lahore, Rawalpindi, Multan, Peshawar and Quetta.

Sample Size:

A total of 90 individuals (45 in each arm) meeting the eligibility criteria will be recruited to participate in the study from different psychiatric units.

Randomization Participants will be randomized into one of the two treatment conditions (LTP Plus or TAU) through computer generated algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual-V (DSM-V) diagnosed first episode psychosis, schizophrenia, schizoaffective disorder, psychosis not otherwise specified or schizophreniform disorder.
* Parents (Mother or Father), age 18 year and above
* Parents (Mother or Father) having a child from birth to 36 months
* Parents (Mother or Father) living within the catchment area of recruitment site.
* Competent and willing to give informed consent
* Parents (Mother or Father) are stable on medication for at least 3 months prior to the intervention.

Exclusion Criteria:

* Violation of any inclusion criteria
* Failure to perform screening or baseline examinations.
* Patients who will meet the criteria for a DSM-V diagnosis of alcohol or substance abuse (other than for nicotine) within the last month or the criteria for DSM-V alcohol or substance dependence (other than for nicotine) within the last 6 months
* Temporary resident unlikely to be available for follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Change in numbers from first month of recruitment to last month of recruitment (total recruitment period is 12 months)
  The number of parent-child dyads referred by the community health workers/treating psychiatrists, the parents who consented from all eligible parent-child dyads
Attrition Rate | Change in numbers from first month of randomisation to last month of outcome assessments (total time period is 18 months).
  The number participants withdrawn out of those consented to participate
Intervention attendance log | number of sessions attended by each participant in 12 month time
  This log will be maintained to assess the acceptability of the intervention is defined as "the extent participant receiving the intervention consider it to be appropriate"

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale | Change in scores from baseline to 3-month post-randomisation
  This is a structured clinical interview consisting of 30 items designed to assess severity of symptoms over the past week on a 7-point scale. Higher score indicates more severe psychopathology.
Psychotic Rating Scale | Change in scores from baseline to 3-month post-randomisation
  This scale rates features such as frequency, intensity, and interference of hallucinations and delusions on a 4-point scale. Higher score indicates more severe psychopathology.
Parenting Stress Index | Change in scores from baseline to 3-month post-randomisation
  This is a a five-point scale to assess (1) Parenting Distress, (2) Difficult Child Characteristics, and (3) Dysfunctional Parent-Child Interaction. Higher score indicates higher intensity of parenting stress.
Maternal Attachment Inventory | Change in scores from baseline to 3-month post-randomisation
  A 26-item scale will be used to ask respondents to indicate how they generally feel in relation to thoughts (e.g. 'My thoughts are full of my baby'), feelings (e.g. 'I feel love for my baby') and situations (e.g. 'I watch my baby sleep') new mothers may experience. Higer score indicate greater level of maternal attachment.
Knowledge attitude and practices of Child Development | Change in scores from baseline to 3-month post-randomisation
  A 20-item questionnaire will be used to assess maternal knowledge and expectations for child development in the first three years. Higher score indicate better knowledge about child development.
Calgary Depression Scale | Change in scores from baseline to 3-month post-randomisation
  This is a depression rating scale especially developed for assessing depression in schizophrenia. Higher scores indicate higher depressive symptom severity.
Social and Occupational Functioning Scale | Change in scores from baseline to 3-month post-randomisation
  It is a global rating of current functioning; this instrument focuses on social and occupational functioning that is independent of the overall severity of the individual's psychological symptoms. Higher score indicate better functioning.
Euro-Qol 5 Dimensions | Change in scores from baseline to 3-month post-randomisation
  A standardized tool assessing the five health related quality of life aspects such as mobility, self-care, typical activates, pain and discomfort and anxiety/depression. Higher score indicate better quality of life.
Client Service Receipt Inventory | Change in scores from baseline to 3-month post-randomisation
  this instrument is used to gather information about the complete spectrum of services and assistance that study participants might utilize
Ages and Stages Questionnaire | Change in scores from baseline to 3-month post-randomisation
  parent-reported screening instrument comprising of 25/29 items focusing social and emotional challenges, Higher score indicate better development.
Manchester Assessment of Caregiver-Infant Interaction | Change in scores from baseline to 3-month post-randomisation
  Six-minute videos of caregiver-infant interaction will be evaluated for a subset of participants by a trained, reliable rater on 7 MACI scales which globally assess core characteristics of caregiver-infant play interaction on a 7-point scale. Higher score indicate better interaction.
Bayley Scale of infant development | Change in scores from baseline to 3-month post-randomisation
  Bayley Scale will be administered on a subset of participants to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infant and toddlers, ages 0-3. Higher score indicate better development.
Child Height | Change in scores from baseline to 3-month post-randomisation
  Child height will be assessed in centimetres
Child Weight | Change in scores from baseline to 3-month post-randomisation
  Child weight will be assessed in KGs
Child head circumference | Change in scores from baseline to 3-month post-randomisation
  This will be assessed in centimetres

CONTACTS AND LOCATIONS:
Locations (1):
- Karwan e hayat, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Only anonymised data will be shared with other researchers ona reasonable request to key contact person.
Supporting Information: Study Protocol
Time Frame: After publication of the trial main results
Access Criteria: Email to corresponding author

REFERENCES:
- [Result] Husain N, Kiran T, Fatima B, Chaudhry IB, Husain M, Shah S, Bassett P, Cohen N, Jafri F, Naeem S, Zadeh Z, Roberts C, Rahman A, Naeem F, Husain MI, Chaudhry N. An integrated parenting intervention for maternal depression and child development in a low-resource setting: Cluster randomized controlled trial. Depress Anxiety. 2021 Sep;38(9):925-939. doi: 10.1002/da.23169. Epub 2021 May 19. PMID 34010505
- [Result] Husain N, Zulqernain F, Carter LA, Chaudhry IB, Fatima B, Kiran T, Chaudhry N, Naeem S, Jafri F, Lunat F, Haq SU, Husain M, Roberts C, Naeem F, Rahman A. Treatment of maternal depression in urban slums of Karachi, Pakistan: A randomized controlled trial (RCT) of an integrated maternal psychological and early child development intervention. Asian J Psychiatr. 2017 Oct;29:63-70. doi: 10.1016/j.ajp.2017.03.010. Epub 2017 Mar 21. PMID 29061430
- [Result] Husain MI, Chaudhry IB, Khoso AB, Wan MW, Kiran T, Shiri T, Chaudhry N, Mehmood N, Jafri SF, Naeem F, Husain N. A Group Parenting Intervention for Depressed Fathers (LTP + Dads): A Feasibility Study from Pakistan. Children (Basel). 2021 Jan 6;8(1):26. doi: 10.3390/children8010026. PMID 33419080
- [Result] Husain MO, Chaudhry IB, Mehmood N, Rehman RU, Kazmi A, Hamirani M, Kiran T, Bukhsh A, Bassett P, Husain MI, Naeem F, Husain N. Pilot randomised controlled trial of culturally adapted cognitive behavior therapy for psychosis (CaCBTp) in Pakistan. BMC Health Serv Res. 2017 Dec 6;17(1):808. doi: 10.1186/s12913-017-2740-z. PMID 29207980